CLINICAL TRIAL: NCT01583829
Title: Randomized Control Trial of Two Computer-Based Attention Training Programs in Schools for Children With Attention Deficit/Hyperactivity Disorder (ADHD)
Brief Title: Study of Computer Attention Training Programs in Schools for Children With Attention Deficit/Hyperactivity Disorder
Acronym: CATS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tufts Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 8926
Record Dates: First submitted 2012-04-16; First posted 2012-04-24 (Estimated); Last update posted 2017-07-07 (Actual); Status verified 2017-07

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: ADHD; neurofeedback; biofeedback; computer attention training
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Neurofeedback; Cognitive Training

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Neurofeedback (Experimental)
  Interventions: Behavioral: Neurofeedback
- Cognitive Training (Experimental)
  Interventions: Behavioral: Cognitive Training
- Waitlist Control (Active Comparator)
  Interventions: Other: Waitlist Control

INTERVENTIONS:
Behavioral: Neurofeedback — 3 times per week for 45 minutes for a total of 40 sessions
  Arms: Neurofeedback
Behavioral: Cognitive Training — 3 times per week for 45 minutes for a total of 40 sessions
  Arms: Cognitive Training
Other: Waitlist Control — 6 30 minute calm breathing sessions over the course of 4 months
  Arms: Waitlist Control

SUMMARY:
This study examines the efficacy of two computer-based attention training systems, one with and one without neurofeedback. The training systems intend to help children learn to focus and attend more effectively.

DETAILED DESCRIPTION:
The current study is examining a neurofeedback (NF) computer attention training system that teaches children to alter their brainwave activity with a Cognitive Training attention training system (CT). The investigators hypothesize that both treatments will show improvement in ADHD symptoms and academic outcomes compared to a control condition.

104 children with ADHD in grades 2 and 4 are randomly assigned to receive the NF, CT, or a Waitlist-Control (WLC) condition that receives NF or CT the following academic year. Children receive forty 45-minute sessions three times a week at school for 4 months. A comprehensive assessment, consists of data completed by teachers, parents, participants, and double-blind classroom observations.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of ADHD (any subtype, per report of the child's physician or school psychologist) entering 2nd or 4th grade at the beginning of September 2009 and 2010.
* combined IQ (Intelligence Quotient) at or above 80,
* ability to read English sufficiently to complete assessments and intervention protocols

Exclusion Criteria:

* mental retardation,
* coexisting diagnosis of conduct disorder,
* pervasive developmental disorder, or
* other serious mental illness (eg., bipolar disorder, psychosis, autism)

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 104 (Actual)
Dates: Start 2009-05; Primary Completion 2012-12 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Behavioral Observations of Students in School (BOSS) | up to three years
  For the purpose of this study, the BOSS is a double blind classroom observation. Each participant is observed by a trained researcher for 15 minutes three times over the course of two days at each assessment point (before the intervention, after the intervention, and at a 6-month follow up) and is evaluated in the areas of off task behaviors (motor, verbal, and passive) and on task behaviors (active and passive).

CONTACTS AND LOCATIONS:
Overall Officials: Naomi J Steiner, MD, Principal Investigator — Tufts Medical Center
Locations (1):
- Tufts Medical Center, Boston, Massachusetts, United States